CLINICAL TRIAL: NCT03373643
Title: Association Between Obstructive Sleep Apnea and Non-alcoholic Fatty Liver Disease Investigated by Liver Biopsy
Brief Title: Obstructive Sleep Apnea and Non-alcoholic Fatty Liver Disease
Acronym: NASHSAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UHAngers
Record Dates: First submitted 2017-11-13; First posted 2017-12-14 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Non-alcoholic Fatty Liver Disease; Sleep Apnea, Obstructive
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient suspected for NAFLD (Experimental)
  Interventions: Diagnostic Test: OSA screening

INTERVENTIONS:
Diagnostic Test: OSA screening — Full night polysomnography

SUMMARY:
Obstructive sleep apnea (OSA) and nonalcoholic fatty liver disease (NAFLD) are frequently encountered in patients with metabolic syndrome (MS). Several data suggest that OSA per se could be a risk factor of liver injury. Most previous studies evaluating the association between OSA severity and the severity of NAFLD used indirect markers of NAFLD including liver imaging or liver injury blood markers or have been performed in morbidly obese patients undergoing intraoperative needle liver biopsy during bariatric surgery.

The current study propose to investigate with a full night polysomnography consecutive patients undergoing percutaneous liver biopsy for suspected NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Suspected NAFLD requiring per-cutaneous liver biopsy

Exclusion Criteria:

* Other than NAFLD liver disease
* Previously diagnosed or treated OSA
* Excessive alcohol consumption (>220 gr/week for men, >140 gr/week for women)
* Pregnancy
* Surgical treatment for obesity past history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2019-12-14 (Estimated); Study Completion 2020-03-14 (Estimated)

PRIMARY OUTCOMES:
Association between OSA severity marker (apnea hypopnea index per hour on the polysomnography) and significant liver fibrosis (score F3 and F4 of the histological nonalcoholic steatohepatitis [NASH]-CRN classification) | The polysomnography will be performed no more than 3 months after the liver biopsy.
  Apnea hypopnea index per hour of sleep is investigated in each participant using full night polysomnography.
  Significant liver fibrosis will be considered if histological analysis conclude to a fibrosis score of 3 or more using the NASH-CRN classification (F3 and F4).

SECONDARY OUTCOMES:
Association between OSA severity marker (apnea hypopnea index per hour on the polysomnography) and significant nonalcoholic steatohepatitis (3 positive criteria on NASH-CRN classification) | The polysomnography will be performed no more than 3 months after the liver biopsy.
  Apnea hypopnea index per hour of sleep is investigated in each participant using full night polysomnography.
  Significant nonalcoholic steatohepatitis will be considered if histological analysis meets 3 positive criteria on NASH-CRN classification: steatosis score ≥ 1 and lobular inflammation score ≥ 1 and hepatocyte ballooning score ≥ 1.
Association between OSA severity marker (apnea hypopnea index per hour on the polysomnography) and significant liver steatosis (histological steatosis > 33% or stade 2 or more on NASH-CRN) | The polysomnography will be performed no more than 3 months after the liver biopsy.
  Apnea hypopnea index per hour of sleep is investigated in each participant using full night polysomnography.
  Significant liver steatosis will be considered if histological analysis conclude to a histological steatosis of 30% or more or a stade 2 steatosis or more using the NASH-CRN classification.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, Please Select, France

IPD SHARING:
Plan to Share IPD: Undecided